CLINICAL TRIAL: NCT00804219
Title: Characterization of Humoral and Cellular Immunity of Low and High-responders After TBE Vaccination
Brief Title: Humoral and Cellular Immunity of Low and High-responders After Tick-borne Encephalitis Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Ursula Wiedermann-Schmidt, Institute of Specific Prophylaxis and Tropical Medicine, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FSME low-responder 1.1; EK Nr 474/2008 (Other: Ethics comitee, Medical University Vienna)
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-11

CONDITIONS: Tick-borne Encephalitis
Keywords: low responsiveness after vaccination
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Influenza Vaccines

ARMS (3):
- TBE low responder (Experimental)
  Interventions: Biological: TBE vaccination and influenza vaccination
- FSME responder (Experimental)
  Interventions: Biological: TBE vaccination and influenza vaccination
- hepatitis B non-responder (Experimental)
  Interventions: Biological: TBE vaccination and influenza vaccination

INTERVENTIONS:
Biological: TBE vaccination and influenza vaccination — FSME-Immun, 0,5 ml, i.m., 1x Inflexal 0,5 ml, i.m., 1x
  Other Names: FSME-Immun ATC code: J07 BA1; Inflexal ATC code: J07 BB02

SUMMARY:
The phenomenon of no- and low-responsiveness has been described after applications of different vaccines (e.g. hepatitis B, TBE) and is concerning about 2-10% of the vaccinees.

The aim of this project is to investigate the humoral and cellular immune responses of low-responders after TBE vaccination in order to find parameters regarding immunoregulation against TBE. It is of interest if non-responsiveness is a general immunological deficit of a distinct patient group or if it is a antigen-specific phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) of both sexes without upper age limit
* Willingness to sign written informed consent form
* Basic vaccination plus one booster (minimum) of TBE-vaccine,

Exclusion Criteria:

* Age: < 18 years
* Pregnancy or breast feeding
* Prior TBE infection
* Planned surgery within 2 weeks before/after any scheduled rabies vaccination during the entire study
* Concomitant medication: systemic cortisone, immune suppressive therapy 4 weeks before or planned medication during the study
* History of autoimmune disease
* Drug addiction
* Plasma donators
* Administration of other vaccines 4 weeks before/after day 0
* Administration of immunoglobulins 6 weeks prior to any vaccination or blood donation during the entire study period
* Specific Immune Therapy (Hypo-/Desensibilization) within 14 days before and after the 2 study vaccination doses.
* History of any malignant disease 5 years prior to the study entry
* Any contraindication for the administration of the TBE- or influenza vaccine according to the manufactures information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
cellular TBE immunity (cytokine production) 7 days after TBE-booster plus influenza vaccination | 7 days after TBE-booster plus influenza vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann-Schmidt, MD, PhD, Principal Investigator — Institute of Specific Prophylaxis and Tropical Medicine
Locations (1):
- Institute of Specific Prophylaxis and Tropical Medicine, Vienna, Vienna, Austria